CLINICAL TRIAL: NCT00709735
Title: A Psychophysiologic Study of Weakening Traumatic Combat Memories With Post-Reactivation Propranolol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Roger K. Pitman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH-07-1-0440
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: stress disorders; post-traumatic; memory; propranolol; psychophysiology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reactivation Propranolol (RP) (Experimental): 0.67 mg/kg short-acting placebo capsules then 1 mg/kg long-acting placebo capsules 90 minutes later on Day 0 (non-reactivation) followed by 0.67 mg/kg short-acting propranolol capsules then 1 mg/kg long-acting propranolol capsules 90 minutes later on Day 2 (reactivation). All participants then underwent a "script preparation" session in which the investigator elicited five discrete personal memories, including two traumatic combat experiences.
  Interventions: Drug: Propranolol; Drug: Placebo
- Non-Reactivation Propranolol (NRP) (Active Comparator): 0.67 mg/kg short-acting propranolol capsules then 1 mg/kg long-acting propranolol capsules 90 minutes later on Day 0 (non-reactivation) followed by 0.67 mg/kg short-acting placebo capsules then 1 mg/kg long-acting placebo capsules 90 minutes later on Day 2 (reactivation). All participants then underwent a "script preparation" session in which the investigator elicited five discrete personal memories, including two traumatic combat experiences.
  Interventions: Drug: Propranolol; Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — 0.67 mg/kg short-acting propranolol combined with 1 mg/kg long-acting propranolol
  Other Names: Inderal
Drug: Placebo — Placebo (matching propranolol) short-acting and long-acting capsules

SUMMARY:
The consolidation of learning is enhanced by adrenalin and other stress hormones. This memory enhancing effect is opposed by propranolol. In posttraumatic stress disorder (PTSD), a psychologically traumatic event may overstimulate stress hormones such as adrenalin, which in turn overly strengthen consolidation of the memory of the event, leading to an excessively powerful and persistent memory. Administration of propranolol after a psychologically traumatic event could reduce subsequent PTSD. Unfortunately, there exists a window of opportunity for influencing the consolidation of a traumatic event into long-term memory. In persons who have already developed PTSD, this would have closed months or years earlier. However, recent developments in animal research suggest that reactivation (retrieval) of a consolidated memory can return it to a labile state, from which it must be restabilized in order to persist. This process, which has been termed "reconsolidation," can be reduced in animals by propranolol.

In a preliminary study performed by the PI and colleagues in Canada, civilian participants with PTSD described the traumatic event during a script preparation session, which served to reactivate their traumatic memory. They then received either propranolol or placebo. A week later, during script-driven imagery of their traumatic events, physiologic responses were smaller in the participants who had received post-reactivation propranolol compared to placebo, suggesting that the traumatic memory had been weakened by the propranolol. These results suggest that that post-reactivation propranolol recapitulates its effects on consolidation, this time by blocking reconsolidation of the traumatic memory.

Several important questions remain unanswered. First, does propranolol also weaken traumatic memories in combat-related PTSD? Second, does this weakening effect only occur when the propranolol is given after combat memory reactivation? If not, this would refute the reconsolidation hypothesis and suggest that propranolol affects non-specific mechanisms. Third, how long does the traumatic memory weakening last?

The proposed project will investigate these questions by performing an improved, double-blind, placebo-controlled study in Iraq and Afghanistan veterans with combat-related PTSD. Participants will be randomly assigned to one of two groups: post-reactivation propranolol or non-reactivation propranolol. Participants in the non-reactivation propranolol group will receive propranolol in the absence of traumatic memory reactivation. Participants randomized to the post-reactivation propranolol group will receive matching placebo capsules. Two days later, all participants will return for a script preparation session, at which time they will describe the details of their traumatic event. Participants randomized to the post-reactivation propranolol group will then receive propranolol, whereas participants randomized to the non-reactivation propranolol group will receive placebo. Participants will then return for psychophysiologic script-driven imagery testing one week and six months later. We hypothesize that those who receive propranolol after reactivation of their memories of their traumatic combat event(s) will show significantly smaller psychophysiologic responses during script-driven imagery testing compared to participants who receive propranolol in the absence of combat memory reactivation, supporting the inference that post-reactivation propranolol blocks the reconsolidation of traumatic combat memories.

DETAILED DESCRIPTION:
Background: Animal evidence indicates that some consolidated memories when reactivated (retrieved) need to be reconsolidated. During this process, memories can be enhanced or weakened. In a preliminary, randomized, double-blind, placebo-controlled study, we tested whether post-reactivation administration of the beta-adrenergic blocker propranolol, which reduces reconsolidation of aversive memories in rodents, would reduce the emotional strength of traumatic memories, or conditioned fear responses, in patients with non-combat-related PTSD. Civilian participants described their traumatic event during a "script preparation" session and thereafter received either a combined dose of short- and long-acting propranolol (n=9), or placebo (n=10). A week later, they engaged in script-driven mental imagery of their personal traumatic events, while peripheral physiologic responses were recorded as measures of the emotional strength of the traumatic memory. We found that physiologic responses were significantly smaller in the participants who had received post-reactivation propranolol compared to placebo a week earlier: F(3,15)=5.1, p=.007, η2=.49. The results of this preliminary study are consistent with pharmacologic blockade of reconsolidation of traumatic memories in PTSD. However, several important questions remain unanswered. First, does propranolol also weaken traumatic memories in combat-related PTSD? Second, does this weakening effect only occur when the propranolol is given when combined with traumatic memory reactivation? If not, this would refute the reconsolidation hypothesis and suggest that propranolol affects non-specific mechanisms. Third, how long does the traumatic memory weakening last, i.e., does recovery of the conditioned fear response occur?

Objective/Hypothesis: The first objective is to replicate and extend the finding from the preliminary study to Iraq and Afghanistan combat veterans with PTSD by showing that propranolol following combat memory reactivation results in a significantly greater weakening of traumatic combat memories than propranolol alone, supporting the proposition that this weakening is due to pharmacological blockade of memory reconsolidation, rather than non-specific actions of propranolol. We hypothesize that participants who undergo script preparation for the combat event(s) that caused their PTSD, followed by (post-reactivation) propranolol, will show significantly smaller psychophysiologic responses during script-driven imagery testing a week later compared to those who receive (non-reactivation) propranolol two days prior to combat script preparation. The second objective to show that this effect is long-lasting, which would be expected if the underlying mechanism is reduction of the traumatic memory trace by blockade of reconsolidation. We hypothesize that the effect will remain significant when participants undergo follow-up psychophysiologic script-driven imagery testing six months later.

Specific Aim: To perform a controlled, randomized, double-blind study in Iraq and Afghanistan veterans with combat-related PTSD that addresses the above hypotheses.

Study Design: Participants will be randomly assigned to one of two groups: post-reactivation propranolol or non-reactivation propranolol. After written informed consent is obtained, participants randomized to the non-reactivation propranolol group will receive a "test" dose of 0.67 mg/kg short-acting propranolol combined with 1 mg/kg long-acting propranolol. Participants randomized to the post-reactivation propranolol group will receive matching placebo capsules. Two days later, all participants will return for an approximate 15-30 minute "script preparation" session, at which time they will describe the details of their traumatic combat event(s) to the Principal Investigator. Participants randomized to the post-reactivation propranolol group will then receive the combined propranolol dose, whereas participants randomized to the non-reactivation propranolol group will receive placebo. Based upon the history obtained during the script preparation session, the Principal Investigator will compose "scripts" approximately 30 seconds in duration portraying each participant's combat events in their own words. Participants will then return for script-driven imagery testing sessions in the psychophysiology laboratory one week and six months later. During each of these sessions, they will undergo recording of heart rate, skin conductance, and corrugator and frontalis electromyogram during a baseline period. They will then listen to a recording of their traumatic scripts and be instructed to imagine the events portrayed as if they were happening again, while physiologic measures are recorded. Responses (change) scores for each physiologic variable for each session will be calculated by subtracting the preceding baseline period mean from the imagery period mean. The physiologic data will be analyzed by multivariate analysis of variance (MANOVA) followed by univariate ANOVAs. The hypothesis predicts that at each time period, the physiologic responses of the post-reactivation propranolol group will be significantly smaller than those of the non-reactivation propranolol group.

Relevance: If a traumatic memory undergoes reconsolidation when reactivated, this could re-open the window of opportunity to influence the memory pharmacologically. This could have important implications for the treatment of PTSD. Should the proposed psychophysiologic study confirm that post-reactivation propranolol weakens traumatic combat memories, it would be a relatively short leap to clinical studies of the therapeutic efficacy of this novel modality.

ELIGIBILITY:
Inclusion Criteria: Afghanistan and Iraq War veterans who have been diagnosed as having combat-related PTSD

Exclusion Criteria:

1. PTSD Checklist (PCL) score (administered at the referring site) ≤ 50;
2. Current, co-existing PTSD of non-combat origin
3. Resting systolic blood pressure <100 mm Hg
4. Medical condition that contraindicates the administration of propranolol
5. Previous adverse reaction to, or non-compliance with, a β-adrenergic blocker
6. Presence of drugs of abuse
7. Pregnancy
8. Contraindicating psychiatric condition
9. Initiation of, or change in, psychotropic medication within the two months prior to recruitment
10. Current use of medication that may involve potentially dangerous interactions with propranolol
11. Inability to understand the study's procedures, risks, and side effects, or to otherwise give informed consent for participation
12. Does not understand English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Pitman, M.D., Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - VA Medical Center, Bedford, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - VA Medical Center, Manchester, New Hampshire

REFERENCES:
- [Result] Wood NE, Rosasco ML, Suris AM, Spring JD, Marin MF, Lasko NB, Goetz JM, Fischer AM, Orr SP, Pitman RK. Pharmacological blockade of memory reconsolidation in posttraumatic stress disorder: three negative psychophysiological studies. Psychiatry Res. 2015 Jan 30;225(1-2):31-39. doi: 10.1016/j.psychres.2014.09.005. Epub 2014 Sep 16. PMID 25441015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Reactivation Propranolol (NRP) | Reactivation Propranolol (RP)
Started | 11 | 12
Completed | 8 | 10
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Relapse into Opioid Abuse | 0 | 1
Not completed — Did not meet PTSD Diagnostic Criteria | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Reactivation Propranolol (NRP) | Reactivation Propranolol (RP) | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (11.5) | 38.7 (14.9) | 36.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 10 | 18
Clinician-Administered PTSD Scale (CAPS) Score [Mean (Standard Deviation); unit: score on a scale] — The clinician evaluated the overall frequency and intensity/severity of the participant's PTSD symptoms using the CAPS. 17 Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) PTSD symptoms were assessed using a 5-point scale for intensity where 0=none to 4=extreme and a 5-point scale for frequency where 0=never to 4=most or all of the time. The intensity score and the frequency scores were added together for a total possible score of 0 (best) to 136 (worst).
  score on a scale | 58.6 (14.8) | 62.7 (13.7) | 60.9 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Physiological Posterior Probability of Posttraumatic Stress Disorder (PTSD) as Determined From Psychophysiologic Responses During Script-Driven Traumatic Memory Recollection
Description: The posterior probability of developing PTSD was determined for each participant from a composite of psychophysiological responses during script-driven imagery of traumatic combat events that included assessments of heart rate response in beats per minute, skin conductance response in microSiemens, and corrugator and left lateral frontalis facial muscle electromyogram (EMG) responses in microVolts. Responses for the two traumatic scripts were averaged and square-root transformed for analysis. Responses during personal traumatic imagery of previously studied individuals with and without current PTSD was used to calculate each participant's posterior probability of being classified as PTSD.
Time Frame: Day 8
Population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: percent probability
Arm/Group | Non-Reactivation Propranolol (NRP) | Reactivation Propranolol (RP)
Number analyzed (Participants) | 8 | 10
percent probability | 32 (11) | 45 (21)
Statistical Analysis 1: Comparison: Non-Reactivation Propranolol (NRP) vs Reactivation Propranolol (RP); Test type: Superiority; Mean Difference (Final Values) = -13.0, 95% CI 2-sided [-30.0 to 4.0] — Non-Reactivation Propranolol (NRP) - Reactivation Propranolol (RP)

2. Secondary Outcome: Change From Baseline in the Impact of Event Scale-Revised (IES-R) Total Score
Description: IES-R is a 22-item patient reported measure of PTSD symptoms. Each question is answered using a 5-point scale where 0=not at all to 4=extremely for a total possible score of 0 to 88. Lower scores represent less severe symptoms and higher scores representing more severe symptoms. IES-R change scores were calculated by subtracting the Day 2 IES-R total score from the Day 8 IES-R total score. A negative change from Baseline indicates improvement of symptoms and a positive change from Baseline indicates a worsening of symptoms.
Time Frame: Day 2 (Baseline ) and Day 8
Population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Reactivation Propranolol (NRP) | Reactivation Propranolol (RP)
Number analyzed (Participants) | 8 | 10
score on a scale
  Baseline | 43.3 (14.2) | 45.0 (18.3)
  Change from Baseline at Day 8 | -8.2 (13.0) | 4.5 (13.2)
Statistical Analysis 1: Comparison: Non-Reactivation Propranolol (NRP) vs Reactivation Propranolol (RP); Test type: Superiority; Mean Difference (Final Values) = -12.7, 95% CI 2-sided [-27.4 to 1.9] — Non-Reactivation Propranolol (NRP) - Reactivation Propranolol (RP)

ADVERSE EVENTS:
Description: All randomized participants who received study drug,
Arm/Group | Non-Reactivation Propranolol (NRP) | Reactivation Propranolol (RP)
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Reactivation Propranolol (NRP) (N=11) | Reactivation Propranolol (RP) (N=12)
Relapse of substance abuse (Psychiatric disorders) | 0 (0) | 1 (1) — One participant in the RP group was withdrawn from the study following his relapse into opioid abuse following his Day 2 participation. This relapse was attributed to the stress of narrating his traumatic event.

LIMITATIONS AND CAVEATS:
Small participant sample due to recruitment difficulties.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No